CLINICAL TRIAL: NCT03064685
Title: Risk Factors and Outcomes of Pyogenic Liver Abscess in Adult Liver Recipients: A Match Case Control Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, Clinical Professor, Hospital Italiano de Buenos Aires
Other Study IDs: 3087
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Liver Transplant Abscess
Keywords: Pyogenic Liver abscess; Liver transplantation; Biliary disease
MeSH Terms: conditions — Liver Abscess, Pyogenic; Gallbladder Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I - Cases: Patients older than 18 years of age with a history of liver transplantation since January 2002 for any cause and who have undergone medical follow-up at HIBA and had at least one event of pyogenic liver abscess after transplantation.
- Group II - Controls: Patients older than 18 years with a history of liver transplantation since January 2002 for any cause and who have performed their medical follow-up at HIBA without developing any event of pyogenic liver abscess after transplantation

SUMMARY:
Objective: the aim of this study is to identify risk factors associated with the development of pyogenic liver abscesses (PLA) in adult liver recipients (ALR) and to describe the experience of the Hospital Italiano de Buenos Aires (HIBA) in the diagnosis and therapeutic management of these patients.

Background: adult liver recipients differ from the general population with PLA as they exhibit: reconstructed biliary anatomy, recurrent hospitalizations, regular performance status and are subjected to immunosuppression. However, the scientific evidence regarding PLA developed in transplanted organs is still scarce and the management of this disease continues to be based on experience in non-transplanted patients.

Methods: between 1996 and 2016, 879 adult patients underwent liver transplantation (LT) at our institution. Patients who developed PLA after LT (cases) and controls are matched according to the time from transplant to abscess in a 1 to 5 relation. The investigators performed a logistic regression model to establish PLA risk factors considering clusters for matched cases and controls. Independent risk factors will be identified using multivariate regression analysis.

DETAILED DESCRIPTION:
Objective: the aim of this study is to identify risk factors associated with the development of pyogenic liver abscesses (PLA) in adult liver recipients (ALR) and to describe the experience of the Hospital Italiano de Buenos Aires (HIBA) in the diagnosis and therapeutic management of these patients.

Background: adult liver recipients differ from the general population with PLA as they exhibit: reconstructed biliary anatomy, recurrent hospitalizations, regular performance status and are subjected to immunosuppression. However, the scientific evidence regarding PLA developed in transplanted organs is still scarce and the management of this disease continues to be based on experience in non-transplanted patients.

Methods: between 1996 and 2016, 879 adult patients underwent liver transplantation (LT) at our institution. Patients who developed PLA after LT (cases) and controls are matched according to the time from transplant to abscess in a 1 to 5 relation. The investigators performed a logistic regression model to establish PLA risk factors considering clusters for matched cases and controls. Independent risk factors will be identified using multivariate regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age with a history of univisceral liver transplantation since January 2002 for any cause and who have undergone medical follow-up at HIBA and had at least one event of liver abscess after transplantation.

Exclusion Criteria:

* Patients who died during the hospitalization of the transplant. Patients with parasitic, fungal or amoebic abscesses were excluded. Those patients with subdiaphragmatic or subhepatic abscesses, tumors with abscessed central necrosis were not included in the study either. Patients who underwent liver transplantation at another institution and were then admitted to hospital with a diagnosis of AHP were not included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years of age with a history of univisceral liver transplantation since January 2002 for any cause and who have undergone medical follow-up at HIBA
Sampling Method: Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2016-11-22 (Actual); Primary Completion 2017-03-02 (Estimated); Study Completion 2017-03-03 (Estimated)

PRIMARY OUTCOMES:
Development of a pyogenic liver abscess after liver transplantation | January 1996 and December 2016
  The diagnosis of hepatic abscess was based on clinical findings, evidence obtained from imaging studies, blood cultures, purulent material obtained from punctures, intraoperative findings and resolution after antibacterial chemotherapy, and one of the following scenarios could be found:
  to. Findings of one or more intrahepatic images of liquid characteristics by means of ultrasound and / or CT scan associated with suspected hepatic abscess based on the clinical picture, laboratory tests and / or microbiological study.
  B. Finding one or more intrahepatic images of liquid characteristics by means of US and / or CT, with posterior drainage of pus.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Peron 4190, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No